CLINICAL TRIAL: NCT04582968
Title: A Phase Ib/II Pilot Study of Pyrotinib Plus Capecitabine Combined With Brain Radiotherapy in HER2 Positive Breast Cancer Patients With Brain Metastases
Brief Title: Pyrotinib Combined With Brain Radiotherapy in Breast Cancer Patients With Brain Metastases
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaoli Yu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-BC010
Record Dates: First submitted 2020-10-07; First posted 2020-10-12 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer; Brain Metastases; HER2-positive Breast Cancer
Keywords: pyrotinib; brain radiotherapy
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib Plus Capecitabine combined with brain radiotherapy (Experimental): Fractionated stereotactic radiotherapy(FSRT) or whole brain radiation therapy (WBRT) Drug: Pyrotinib combined with capecitabine pyrotinib 400 mg once daily; Capecitabine 1000 mg/m2 per day on day 1 through 14, every 21 days.
  Interventions: Other: Pyrotinib Plus Capecitabine combined with brain radiotherapy

INTERVENTIONS:
Other: Pyrotinib Plus Capecitabine combined with brain radiotherapy — Drug combined with radiation

SUMMARY:
Brain metastases occur in 30-50% of patients with metastatic HER2-positive breast cancer. Pyrotinib is an irreversible pan-ErbB receptor tyrosine kinase inhibitor (TKI) with activity against epidermal growth factor receptor (EGFR)/HER1, HER2, and HER4. This study consists of two parts. In a phase Ib part, investigators will explore the safety and tolerance of Pyrotinib Plus Capecitabine combined with brain radiotherapy. After completing the phase Ib part, investigators will review the data and decide whether this patient is included in before the start of a phase II part. In the phase II part, investigators will evaluate the efficacy of Pyrotinib Plus Capecitabine combined with brain radiotherapy in patients with HER2 positive breast cancer patients with brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed HER2 positive advanced breast cancer
2. Age>18 years. brain metastases confirmed by enhanced brain MRI
3. KPS≥70
4. Life expectancy of more than 12 weeks
5. Prior therapy of oral dexamethasone not exceeding 16mg/d
6. Time interval from prior therapy was more than 2 weeks, and evaluation of adverse events is no more than grade 1.
7. Maximum diameter of intracranial metastases is less than 3cm measured by enhanced brain MRI(2-3mm)
8. Prior endocrine therapy were allowed
9. Anti-Her2 targeted treatment were allowed
10. Screening laboratory values must meet the following criteria( and should be obtained within 28 days prior to registration):

    1. Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L, Platelets≥ 90 x 109/L, Hemoglobin ≥ 90 g/L
    2. Aspartate aminotransferase/alanine aminotransferase (AST/ALT) ≤2.5 x ULN without liver metastasis,≤ 5 x ULN with liver metastases
    3. Serum BUN and creatinine ≤ 1.5 x Upper Limit of Normal (ULN)
    4. LVEF ≥ 50%
    5. QTcF < 480 ms
    6. INR≤1.5×ULN，APTT≤1.5×ULN
11. Signed the informed consent form prior to patient entry

Exclusion Criteria:

1. Leptomeningeal or hemorrhagic metastases
2. uncontrolled epilepsy
3. Severe complication: cardiovascular disease, end-stage renal disease, severe hepatic disease, infection etc.
4. Pregnancy or lactation period， women of child-bearing age who are unwilling to accept contraceptive measures.
5. Inability to complete enhanced MRI
6. Patients who are difficult or unable to be followed-up
7. Not suitable for inclusion for specific reasons judged by sponsor
8. Patients unable to swallow, with chronic diarrhea, intestinal obstruction, or multiple factors that affect drug use and absorption
9. History of allergy to pyrotinib or capetabine
10. History of immunodeficiency, including HIV positive, active HBV/HCV or other acquired, congenital immunodeficiency disease, or organ transplantation history
11. Previous use of pyrotinib combined with capetabine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2023-08-12 (Estimated)

PRIMARY OUTCOMES:
Assess safety and tolerability of Pyrotinib Plus Capecitabine combined with brain radiotherapy(Phase Ib part) | 8 weeks
  AEs will be assessed according to CTCAE version 4.03.
  (1)Initially 3 patients will be accrued and treated with combined therapy as a lead-in safety phase. Enrollment of the study will not proceed if patients in the safety lead-in phase experience unacceptable toxicities including neurologic, hematologic and other dose limiting toxicities.(see protocol) (b)If one of initially 3 patients has experienced unacceptable toxicities, 3 more patients will be accrued .
  (3)If two or more patients are unable to complete radiation therapy (RT) due to toxicity related to Pyrotinib Plus Capecitabine combined with brain radiotherapy, accrual will be suspended and the study will be stopped.
  (4) If 3+3 patients are able to complete the treatment without unacceptable toxicities, 6 more patients will be accrued in Ib part.
Intracranial local tumor control rate （Phase II part) | 2 years
  All intracranial progression

SECONDARY OUTCOMES:
Intracranial local tumor control rate with FSRT or WBRT | 2 years
  Intracranial local tumor control rate
Intracranial Progression-Free Survival (PFS) | 2 years
  Time from the date of radiotherapy to the investigator-determined date of progression (determined by RANO) or death due to any cause, whichever occurs first
Extracranial Progression-Free Survival (PFS) | 2 years
OS (overall survival) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Yu, MD PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

REFERENCES:
- [Derived] Dai L, Gao T, Guo R, Chen Y, Wang J, Zhou S, Tang Y, Chen D, Huang S. Efficacy and safety of pyrotinib-based regimens in HER2 positive metastatic breast cancer: A retrospective real-world data study. Neoplasia. 2024 Oct;56:101029. doi: 10.1016/j.neo.2024.101029. Epub 2024 Jul 17. PMID 39024777
- [Derived] Yang Z, Meng J, Mei X, Mo M, Xiao Q, Han X, Zhang L, Shi W, Chen X, Ma J, Palmer J, Shao Z, Zhang Z, Yu X, Guo X. Brain Radiotherapy With Pyrotinib and Capecitabine in Patients With ERBB2-Positive Advanced Breast Cancer and Brain Metastases: A Nonrandomized Phase 2 Trial. JAMA Oncol. 2024 Mar 1;10(3):335-341. doi: 10.1001/jamaoncol.2023.5791. PMID 38175627